CLINICAL TRIAL: NCT00905853
Title: Ventricular Tachycardia Ablation or Escalated aNtiarrhythmic Drugs in ISchemic Heart Disease
Brief Title: Ventricular Tachycardia (VT) Ablation or Escalated Drug Therapy
Acronym: VANISH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: John Sapp (Other)
Collaborators: Abbott Medical Devices (Industry); Biosense Webster, Inc. (Industry); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor-Investigator, John Sapp, Staff physician, Division of Cardiology, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sapp001
Record Dates: First submitted 2009-05-20; First posted 2009-05-21 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Recurrent Ventricular Tachycardia
Keywords: Ventricular Tachycardia; Catheter Ablation; ICD therapy; Antiarrhythmic Drug Therapy; Ischemic Heart Disease
MeSH Terms: conditions — Tachycardia, Ventricular; Myocardial Ischemia | interventions — Catheter Ablation; Amiodarone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ventricular Tachycardia Ablation (Active Comparator): Catheter ablation for Ventricular tachycardia will be performed within 14 days of randomization.
  Interventions: Procedure: Catheter Ablation
- Escalated Antiarrhythmic Drug Therapy (Active Comparator): Patients are prescribed a loading dose of amiodarone or the addition of mexiletine to their current anti-arrhythmic medication which is stratified by the dose and type of antiarrhymic medication at the time of the index arrhythmic event.
  Interventions: Drug: Escalated Antiarrhythmic Therapy

INTERVENTIONS:
Procedure: Catheter Ablation — Intracardiac electrode catheters are placed via central vasculature to identify myocardial scar, and surviving conduction channels within the scar which form the substrate for ventricular tachycardia. Radiofrequency energy is applied to these sites, interrupting the VT circuits.
  Other Names: VT Ablation
  Arms: Ventricular Tachycardia Ablation
Drug: Escalated Antiarrhythmic Therapy — Patients who have 'failed' antiarrhythmic therapy (except amiodarone) will be prescribed: Amiodarone 400 mg twice daily for 2 weeks, followed by 400 mg/day for 4 weeks, followed by 200 mg/day thereafter.
  Patients who 'failed' amiodarone (less than 300mg/day) will be prescribed: Amiodarone 400 mg three times a day for 2 weeks, followed by 400 mg/day for 1 week and 300 mg/day thereafter.
  Patients who 'failed' amiodarone (greater or equal to 300mg/day) will be prescribed: Amiodarone at the current dose with the addition of mexiletine 400 to 800 mg/day
  Other Names: Cordarone; Mexetil
  Arms: Escalated Antiarrhythmic Drug Therapy

SUMMARY:
This study will compare aggressive antiarrhythmic therapy to catheter ablation for ventricular tachycardia in patients who have suffered prior myocardial infarction. The purpose of this study is to evaluate the optimal management of patients presenting with recurrent VT and receiving ICD therapy in spite of first-line antiarrhythmic drug therapy. The hypothesis is catheter ablation is superior to aggressive antiarrhythmic drug therapy for recurrent VT.

DETAILED DESCRIPTION:
This is a multicentre, parallel group, two arm, unblinded, randomized clinical trial to compare two management strategies for patients with ischemic heart disease and recurrent ICD therapy despite at least one antiarrhythmic drug. The primary endpoint will be a composite of appropriate ICD shocks or death.

ELIGIBILITY:
Inclusion Criteria:

* Prior Myocardial Infarction
* An implantable defibrillator
* One of the following VT events (within the past 3 months):

  * greater than or equal to 3 episodes of symptomatic VT treated with ATP
  * greater than or equal to 1 appropriate ICD shock
  * greater than or equal to 3 VT episodes within 24 hours
  * sustained VT below detection rate of the ICD documented by ECG
* "Failed" first-line antiarrhythmic drug therapy as defined by one of:

  * Appropriate ICD therapy or sustained VT occurred while patient was taking amiodarone (stable dose >/= 2 weeks)
  * Appropriate ICD therapy or sustained VT occurred on another antiarrhythmic drug (stable dose >/= 2 weeks)

Exclusion Criteria:

* Active ischemia (acute thrombus, dynamic ST elevation on ECG) or another reversible cause of VT (eg. electrolyte abnormalities, drug induced arrhythmia)
* Are known to be ineligible to take amiodarone (eg. active hepatitis, current hyperthyroidism, pulmonary fibrosis, known allergy)
* Are ineligible for ablation (left ventricular thrombus, implanted mechanical aortic and mitral valves)
* Renal Failure (creatinine clearance < 15 ml/min)
* Current NYHA functional class IV heart failure or CCS Functional Class IV angina
* Recent ST elevation myocardial infarction (< 1 month)
* Recent coronary bypass surgery (< 3 mon) or recent PCI (< 1 mon)
* Pregnant
* prior ablation for ventricular tachycardia
* A systemic illness likely to limit survival to < 1 year
* Unable or unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2009-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Appropriate ICD shocks,VT storm and death | 3 years

SECONDARY OUTCOMES:
All cause mortality | 3 years
Appropriate ICD antitachycardia pacing anytime and after 1 month treatment period | 3 years
appropriate ICD shocks anytime and after 1 month treatment period | 3 years
Inappropriate shocks anytime and after 1 month treatment period | 3 years
VT storm anytime and after 1 month treatment period | 3 years
Documented sustained VT below detection rate of the ICD any time and after 1 month treatment period | 3 years
Number of ICD shocks | 3 years
Hospital admission for cardiac causes | 3 years
Procedural complications, amiodarone toxicity or adverse events | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: John L Sapp, BSc, MD, FRCPC, Principal Investigator — Nova Scotia Health Authority; Ratika Parkash, MD, MSc, FRCPC, Study Director — Nova Scotia Health Authority; Anthony S Tang, MSc, MD, FRCPC, Study Director — Royal Jubilee Hospital; George A Wells, BSc,MSc,PhD, Study Director — Univeristy of Ottawa Heart Institute; William G Stevenson, MD, Study Director — Brigham and Women's Hospital
Locations (1):
- QEII Health Sciences Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Parkash R, Nault I, Rivard L, Gula L, Essebag V, Nery P, Tung S, Raymond JM, Sterns L, Doucette S, Wells G, Tang ASL, Stevenson WG, Sapp JL. Effect of Baseline Antiarrhythmic Drug on Outcomes With Ablation in Ischemic Ventricular Tachycardia: A VANISH Substudy (Ventricular Tachycardia Ablation Versus Escalated Antiarrhythmic Drug Therapy in Ischemic Heart Disease). Circ Arrhythm Electrophysiol. 2018 Jan;11(1):e005663. doi: 10.1161/CIRCEP.117.005663. PMID 29305400
- [Derived] Sapp JL, Wells GA, Parkash R, Stevenson WG, Blier L, Sarrazin JF, Thibault B, Rivard L, Gula L, Leong-Sit P, Essebag V, Nery PB, Tung SK, Raymond JM, Sterns LD, Veenhuyzen GD, Healey JS, Redfearn D, Roux JF, Tang AS. Ventricular Tachycardia Ablation versus Escalation of Antiarrhythmic Drugs. N Engl J Med. 2016 Jul 14;375(2):111-21. doi: 10.1056/NEJMoa1513614. Epub 2016 May 5. PMID 27149033